CLINICAL TRIAL: NCT02830620
Title: Study at the Man of the Profile of Chimiokines in the Anorexia Bound to the Cancerous Cachexy.
Acronym: CHIMIOKINES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-PP-03
Record Dates: First submitted 2012-07-20; First posted 2016-07-13 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cancer of the Pancreas; Anorexia
MeSH Terms: conditions — Pancreatic Neoplasms; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- groupe1 (Other): cancer of the pancreas WITH syndrome of anorexia-cachexie Dosage of chimiokines
  Interventions: Other: Dosage of chimiokines
- groupe2 (Other): cancer of the pancreas WITHOUT syndrome of anorexia-cachexie Dosage of chimiokines
  Interventions: Other: Dosage of chimiokines
- groupe3 (Other): pure food limitation typifies restrictive anorexia nervosa Dosage of chimiokines
  Interventions: Other: Dosage of chimiokines
- groupe4 (Other): unhurt individual of any appetite-suppressing evolutionary disease and cachectisante Dosage of chimiokines
  Interventions: Other: Dosage of chimiokines

INTERVENTIONS:
Other: Dosage of chimiokines

SUMMARY:
The syndrome of anorexia-cachexie, which accompanies numerous cancers is a major comorbidity which compromises the forecast of these patients. Several cytokines pro-inflammatory as interleukines IL1 ß, IL6 or TNFa participate in the physiopathology of this syndrome at the man and the animal. Besides, it is now established that different neuronal populations, localized in the hypothalamus, are nerve centers of the control of the appetite and the energy homéostasie. However, there is not enough evidence of a direct action of cytokines on these neurones, suggesting the participation of intermediate molecules as chimiokines, inflammatory molecules produced in reaction to an immunological stress by gliales cells and acting directly on the surrounding neurones. The implication of chimiokines in the syndrome of anorexia-cachexie associated with the cancer thus seems very likely Among these, chimiokines " Monocyte Chemoattractant Proteins 1-3 " or MCPs represent obvious candidates because they are produced by multiple tumors. Furthermore, to the mouse, the intellectual expression of MCP1 is correlated in the anorexia led by peripheral injections of a bacterial by-product, the lipopolysaccharide (LPS).

The investigators' main objective is to test at the Man's, in situation of cancer of the pancreas any confused stages, the degree of prédictivité of the chimiokine MCP1 towards the syndrome of anorexia-cachexie associated with the cancer. The investigator also suggest describing: i) the link between rate plasmatique of MCP1 and energy metabolism on one hand, physical composition on the other hand;; ii) the impact of the other chimiokines, particularly those of the family of the MCPs, on the anorexia-cachexie bound to the cancer, iii) the correlation enters their profile of expression plasmatique and the severity of the anorexia, the energy metabolism and the physical composition; iv) the same research on the other inflammatory factors plasmatiques, of nature different from chimiokines; v) the correlation between thin mass and anorexia; vi) the evolution of the chimiokines various and inflammatory factors after surgical treatment or chemotherapy with curative aim in 6 months.

ELIGIBILITY:
Group 1 {cancer of the pancreas WITH syndrome of anorexia-cachexie}

Inclusion Criteria:

* Patient to hospitalize in the unit of digestive cancer research.
* Patient ≥ 18 years.
* Patient carrier of an adénocarcinome of the pancreas of novo, any stadium confused, diagnosed by imaging and/or histology.
* Existence of at least one of the criteria following to hold(retain) the diagnosis of cachexie cancer patient: not deliberate loss of weight > in 5 % over the last 6 months OR(WHERE) IMC(CEREBRAL-MOTOR HANDICAPPED) < 20 kg / m ² with a loss of minimum weight > 2 % OR(WHERE) scrawny muscular index appendiculaire respectively < 7,26 kg / m ² at the man and < 5,45 kg / m ² at the woman with a minimal weight loss > 2 %.
* Patient having signed the enlightened consent.

Exclusion Criteria:

* Patient having a tumor other one than the pancreatic adénocarcinome.
* Patient having a second offense of adénocarcinome pancreatic.
* Patient carrier of a pancreatic adénocarcinome in the course of a treatment by chemotherapy.
* Patient having a severe psychiatric comorbidity except TCA who can be responsible for food disorders.
* Patient carrier of an evolutionary inflammatory disease other one than the cancer being able to interfere on the inflammatory status.

Groupe 2 {cancer du pancréas SANS syndrome d'anorexie-cachexie}

Inclusion Criteria:

* Patient to hospitalize in the(unit) of digestive cancer research.
* Patient ≥ 18 years.
* Patient carrier of an adénocarcinome of the pancreas of novo, any stadium confused, diagnosed by imaging and/or histology.
* Patient having signed a enlightened consent.

Exclusion Criteria:

* Patient having a tumor other one than the pancreatic adénocarcinome.
* Patient having a second offense(recurrence) of adénocarcinome pancreatic.
* Patient carrier of a pancreatic adénocarcinome in the course of a treatment by chemotherapy.
* Existence of at least one of the criteria in favour of the diagnosis of cachexie cancer patient: not deliberate loss of weight > in 5 % over the last 6 months OR(WHERE) IMC(CEREBRAL-MOTOR HANDICAPPED) < 20 kg / m ² with a loss of minimum weight > 2 % OR(WHERE) scrawny muscular index appendiculaire respectively < 7,26 kg / m ² at the man and < 5,45 kg / m ² at the woman with a minimal weight loss > 2 %.
* Patient having a severe psychiatric comorbidity except TCA who can be responsible for food disorders.
* Patient carrier of an evolutionary inflammatory disease other one than the cancer being able to interfere on the inflammatory status.
* Patient refusing to participate in the study
* Under guardianship patient or guardianship.

Group 3 {pure food limitation typifies restrictive anorexia nervosa}

Inclusion Criteria:

* Patient seen in consultation in the unit of nutritional support(medium)
* Patient ≥ 18 years.
* Patient carrier of an eating disorder of type pure restrictive anorexia nervosa (according to criterion diagnosis of the WHO)
* Patient having signed a enlightened consent.

Exclusion Criteria:

* Patient having any evolutionary organic pathology source of a decrease of the oral contributions and/or the interference on the inflammatory status, and responsible for a loss of weight
* Patient refusing to participate in the study
* Under guardianship patient or guardianship.

Group 4 {unhurt individual of any appetite-suppressing evolutionary disease and cachectisante}

Inclusion Criteria:

* Patient seen in consultation of hepatogastroenterology
* Patient ≥ 18 years.
* Unhurt patient of any organic or psychic, evolutionary pathology, cachectisante
* Patient having signed a enlightened consent.

Exclusion Criteria:

* Patient refusing to participate in the study
* Under guardianship patient or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
chimiokine MCP1 expression | change from baseline to 180 days
  Study at the Man's, in situation of cancer of the pancreas, diagnosed of novo and any confused stages, the prediction of the chimiokine MCP1 towards the syndrome of anorexia-cachexie associated with the cancer

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SCHNEIDER, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France